CLINICAL TRIAL: NCT05931510
Title: Effects of Myofascial Release Versus Post Isometric Relaxation Among Futsal Players With Shin Splints
Brief Title: Release Versus Post Isometric Relaxation Among Futsal Players With Shin Splints
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0425
Record Dates: First submitted 2023-06-26; First posted 2023-07-05 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Shin Splint
Keywords: Shin splint; Myofascial release; Post isometric relaxation
MeSH Terms: conditions — Medial Tibial Stress Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Myofascial release
  Interventions: Other: Myofscual release
- Group B (Experimental): Post isometric relaxation
  Interventions: Other: Post isometric relaxation.

INTERVENTIONS:
Other: Myofscual release — I will apply myofascial release on group A patients and observse its effects on shin splint
  Other Names: Hot pack
  Arms: Group A
Other: Post isometric relaxation. — I will apply post isonetric relaxation on group b patients and observe effects on shin splint
  Other Names: Hot pack
  Arms: Group B

SUMMARY:
The aim of the study is to determine the effects of myofascial release versus post isometric relaxation among futsal players with shin splints

DETAILED DESCRIPTION:
Previous literature did not compare the combined effects of both myofascial release and post isometric relaxation technique inn sgin splints patients so the purpose of this study is self-explanatory, with the basic goal of comparing these two techniques to determine their effects on patient Pain, and Functional disability thus improving overall performance of the futsal players.This study will be helpful in proposing proper treatment for shin splint, to make people aware of the condition rehabilitation and improving performance of the futsal players undergoing the condition. Thus it will be useful for the betterment of the players overall health and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects have leg pain with exertion of more than 1 or 2 hours
* Participants age 20-30 years
* Participants have MTSS for more than 2 weeks
* Subjects have No previous history of trauma to legs
* Subject having Local pain on lower anterior leg Gradual cessation of the offending activity

Exclusion Criteria:

* • Subjects have medical history of systemic disease

  * Subjects have Medical history of cardiovascular disease
  * Participants with History of metastatic diseases
  * Any trauma or pathology of lower limb Participants having Neuropathy of lower extremity

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2022-11-22 (Actual); Primary Completion 2023-07-15 (Estimated); Study Completion 2023-07-25 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 3 months
  Numeric pain rating scale NPRS is a subjective measure in which Pain intensity is frequently measured on an 11-point pain intensity scale (PI-NRS), where 0=no pain and 10=worst possible pain.
Lower extremity functional scale | 3 months
  Lower extremity functional scale LEFS is a valid, reliable, and responsive tool that can be used to measure function in patients with lower extremity musculoskeletal dysfunction

CONTACTS AND LOCATIONS:
Overall Officials: Nosheen Manzoor, Principal Investigator — Riphah International University
Locations (1):
- Model town hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No